CLINICAL TRIAL: NCT01929330
Title: An Evaluation of the Bioequivalence of Five 0.1 mg GI198745/Dutasteride Soft Gelatin Capsules Compared to One 0.5 mg GI198745/Dutasteride Gelatin Capsules in Healthy Male Volunteers
Brief Title: Bioequivalence Study of Dutasteride Five 0.1 mg and One 0.5 mg Soft Gelatin Capsules in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 117342
Record Dates: First submitted 2013-08-22; First posted 2013-08-27 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Alopecia
Keywords: Bioequivalence; Healthy Male Volunteers; Androgenetic Alopecia; Dutasteride; Safety; Tolerability
MeSH Terms: conditions — Alopecia | interventions — Dutasteride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sequence AB (Experimental): Subjects will be hospitalized to the clinical unit on the evening of Day -1. All subjects will receive 1 x 0.5mg oral dose of dutasteride (Sequence A), in the morning; Subjects will remain in the clinical unit until completion of all assessments at 24 hours post-dose on Day 2 including collection of the 24 hour post-dose PK sample. Subjects will return to the unit for the remaining PK samples at 36, 48 and 72 hours. The subject will receive or 5 x 0.1mg oral dose of dutasteride (Sequence B) in similar fashion as that of Sequence A. The two treatment sequences will be separated by a minimum washout period of 28 days to ensure that dutasteride is effectively eliminated from the subject between dosing occasions.
  Interventions: Drug: GI198745 0.1 mg; Drug: GI198745 0.5 mg
- Sequence BA (Experimental): Subjects will be hospitalized to the clinical unit on the evening of Day -1. All subjects will receive 5 x 0.1mg oral dose of dutasteride (Sequence B) in the morning; Subjects will remain in the clinical unit until completion of all assessments at 24 hours post-dose on Day 2 including collection of the 24 hour post-dose PK sample. Subjects will return to the unit for the remaining PK samples at 36, 48 and 72 hours. The subjects will receive 1 x 0.5mg oral dose of dutasteride (Sequence A) in similar fashion as that of Sequence B, The two treatment sequences will be separated by a minimum washout period of 28 days to ensure that dutasteride is effectively eliminated from the subject between dosing occasions.
  Interventions: Drug: GI198745 0.1 mg; Drug: GI198745 0.5 mg

INTERVENTIONS:
Drug: GI198745 0.1 mg — It is available as soft gelatin capsule to be administered as 5 X 0.1 mg capsules as single oral dose with approximately 250 mL of water.
Drug: GI198745 0.5 mg — It is available as soft gelatin capsule to be administered as 1 X 0.5 mg capsules as single oral dose with approximately 250 mL of water.

SUMMARY:
The aim of this study is to determine the bioequivalence of 5 x 0.1 milligram (mg) capsules compared to 1 x 0.5 mg capsule of dutasteride in healthy male subjects. The results of this study are expected to support registration applications for androgenetic alopecia (AGA) in Japan and other international markets.

ELIGIBILITY:
Inclusion Criteria:

* Males aged between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the Investigator, in consultation with the GlaxoSmithKline (GSK) Medical Monitor if required, judges and documents that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Body weight >= 50 kilogram (kg) and body mass index within the range 19 - 32 kg/square meter (m2) (inclusive).
* Male subjects with female partners of child-bearing potential must agree to use a condom. This criterion must be followed from the time of the first dose of study medication until 50 days post last dose.
* Willing and able to give written informed consent, which includes compliance with all the requirements and restrictions listed in the consent form for the full duration of the study, and able to understand and follow instructions related to study procedures.
* Able to swallow and retain oral medication.
* Alanine aminotransferase, Aspartate aminotransferase, alkaline phosphatase and bilirubin <= 2.0 x upper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Based on single or averaged corrected QT interval (QTc) values of triplicate ECGs obtained over a brief recording period: QT duration corrected for heart rate by Fridericia's formula (QTcF) < 450 milliseconds.

Exclusion Criteria:

* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* History of regular alcohol consumption within 6 months of the study defined as:

An average weekly intake of >21 units for males. In Australia one unit (=standard drink) is equivalent to 10 gram of alcohol: 270 milliliter (mL) of full strength beer (4.8%), 375 mL of mid strength beer (3.5%), 470 mL of light beer (2.7%), 250mL pre-mix full strength spirit (5%), 100 mL of wine (13.5%) and 30 mL of spirit (40%).

* History of sensitivity to any of the study medications, or components thereof or a history of drug, or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* History of myocardial infarction, coronary bypass surgery, unstable angina, cardiac arrhythmias, clinically evident congestive heart failure, or cerebrovascular accident prior to Screening visit;
* History of diabetes or peptic ulcer disease which is uncontrolled by medical management.
* History of: Breast cancer or clinical breast examination finding suggestive of malignancy; Malignancy within the past five years, except for basal cell carcinoma of the skin. Subjects with a prior malignancy who have had no evidence of disease for at least the past 5 years are eligible.
* Prior medical history or evidence of prostate cancer (e.g., positive biopsy, or suspicious ultrasound, or suspicious digital rectal examination [DRE]). Patients with suspicious ultrasound or DRE who have had a negative biopsy within the preceding 6 months and stable prostate specific antigen (PSA) are eligible for the study.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* A positive pre-study drug/alcohol screen.
* A positive test for HIV antibody.
* Creatinine >1.5xULN normal
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Unable to refrain from the use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2013-09-23 (Actual); Primary Completion 2014-01-09 (Actual); Study Completion 2014-01-09 (Actual)

PRIMARY OUTCOMES:
Serum pharmacokinetic (PK) parameters: maximum observed concentration (Cmax) and Area under the concentration-time curve from time zero to last time of quantifiable concentration within a subject (AUC[0-t]) for dutasteride | From pre-dose up to 72 hrs
  Serum PK samples will be collected pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 6, 8, 10, 12, 18, 24, 36, 48, and 72 hours post dose for both treatment periods

SECONDARY OUTCOMES:
Time to Cmax (tmax) for dutasteride as data permit | From pre-dose up to 72 hrs
  Serum PK samples will be collected pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 6 8, 10, 12, 18, 24, 36, 48, and 72 hours post dose for both treatment periods
Safety and tolerability of all treatments as assessed by vital signs, electrocardiogram (ECG) measurements, review of adverse events (AEs) and clinical laboratory safety data | From screening till Follow-up visit (10-14 days post-last dose)& 50-54 days post-last dose
  Vital signs will include pulse rate and blood pressure measurements.12-lead ECGs will be obtained at the planned time point. An AE is any untoward medical occurrence temporally associated with the use of the medicinal product, whether or not considered associated with the product. Clinical laboratory tests will include hematology, clinical chemistry and urinalysis parameters.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Randwick, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Fossler MJ, Collins DA, Ino H, Sarai N, Ravindranath R, Bowen CL, Burns O. Evaluation of bioequivalence of five 0.1 mg dutasteride capsules compared to one 0.5 mg dutasteride capsule: a randomized study in healthy male volunteers. J Drug Assess. 2015 Jul 14;4(1):24-9. doi: 10.3109/21556660.2015.1067219. eCollection 2015. PMID 27536459
- See also: Results for study 117342 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/117342?search=study&search_terms=117342#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 117342 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 117342 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 117342 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 117342 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 117342 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 117342 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 117342 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register